CLINICAL TRIAL: NCT06900387
Title: Effect of Oral Vitamin D3 and Calcium Supplementation on Sarcopenia Indices and Osteoporosis Among Rural Post-menopausal Women
Brief Title: Effect of Oral Vitamin D3 and Calcium Supplementation on Muscle and Bone Health Among Rural Post-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Anuradha Khadilkar (Other)
Responsible Party: Sponsor-Investigator, Dr. Anuradha Khadilkar, Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Organization: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JCDC/BHR/23/044
Record Dates: First submitted 2024-12-06; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia; Osteoporosis
Keywords: Sarcopenia intervention study; sarcopenia
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Cholecalciferol; Tablets; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A- Calcium and Vitamin D3 (Active Comparator): Calcium Carbonate tablet (500 mg)- daily for the period of 6 months. Vitamin D3 (Cholecalciferol) tablet (60,000 IU) once a month for the period of 6 months.
  Interventions: Dietary Supplement: Tablet Calcinum-Calcium Carbonate (500mg) daily and Vitamin D3 (Cholecalciferol) tablet (60,000 IU) once a month.
- Group B- Vitamin D3 (Active Comparator): Vitamin D3 (Cholecalciferol) tablet (60,000 IU) once a month for the period of 6 months.
  Interventions: Dietary Supplement: Tablet Tayo- Vitamin D3 (Cholecalciferol) (60,000 IU) once a month.
- Group C- Control Group (Active Comparator): This was a control group. No additional intervention was given to control group.
  Interventions: Other: Control Group

INTERVENTIONS:
Dietary Supplement: Tablet Calcinum-Calcium Carbonate (500mg) daily and Vitamin D3 (Cholecalciferol) tablet (60,000 IU) once a month. — Oral Calcium Carbonate supplement 500 mg from La Renon Healthcare Pvt Ltd to be administered daily for the period of 6 months. Oral Vitamin D3 (Cholecalciferol) supplement 60,000 IU from Eris Lifesciences Ltd to be administered once a month for the period of 6 months.
  Arms: Group A- Calcium and Vitamin D3
Dietary Supplement: Tablet Tayo- Vitamin D3 (Cholecalciferol) (60,000 IU) once a month. — Oral Vitamin D3 (Cholecalciferol) supplement 60,000 IU from Eris Lifesciences Ltd to be administered once a month for the period of 6 months.
  Arms: Group B- Vitamin D3
Other: Control Group — No additional intervention was given to control group.
  Arms: Group C- Control Group

SUMMARY:
This will be three-arm parallel group trial. The goal of this intervention study is to observe the effect of vitamin D3 and calcium supplementation for the period of 6 months on improving the sarcopenia indices such as appendicular muscle mass, muscle strength and muscle function as well as bone density among rural post-menopausal women between age 40 to 65 years. The main questions it aims to answer are:

1. Does the Vitamin D3 supplementation alone help in improving sarcopenia measures or the addition of Calcium supplement along with Vitamin D3 will be more effective in improvement of muscle mass, muscle strength and muscle function.
2. Does Vitamin D3 and Calcium supplementation improve the bone density on supplementation for the period of 6 months among post-menopausal women.

Participants will be given supplementation in three groups in which first group will receive vitamin D3 and calcium supplementation, second group will receive only vitamin D3 supplementation and third group will receive placebo in the form of vitamin B-Complex tablet. Calcium tablet of 500 mg was given daily for the period of 1 month and compliance was checked by collecting empty blisters of tablets from the participants. Vitamin D3 (60,000IU) tablet was given once a month and compliance were checked by observing direct consumption of tablet in front of the care provider/trained social worker. Participants will be measured at the baseline for their muscle and bone parameters and they will visit after 6 months on completion of their supplementation.

Researcher will compare both the supplementation arms (Calcium and vitamin D3 with vitamin D3 alone) with each other and with the third arm of placebo group (supplemented with vitamin B-complex tablet).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy post-menopausal women
2. Age between 40-65 years.

Exclusion Criteria:

1. Women with co-morbidities such as diabetes, thyroid conditions, heart disease, chronic liver/kidney disease, present acute illness
2. Presence of any metal implants in bones
3. Women who have undergone hysterectomy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Sarcopenia Indices | 6 months
  Change in appendicular skeletal muscle index, muscle strength and muscle function in post-menopausal women after supplementation with calcium and vitamin D3 using DXA, JAMAR hand dynamometer and Short Physical Performance Battery
Bone density measures | 6 months
  Change in bone mineral density at lumbar spine and femur neck in post-menopausal women after supplementation with calcium and vitamin D3 using DXA

SECONDARY OUTCOMES:
Vitamin D levels | 6 months.
  Change in Serum vitamin D levels(ng/ml) will be assessed
Parathyroid Hormone (PTH) levels | 6 months
  Change in PTH levels ( pg/ml ) will be assessed
Lipid Profile | 6 months
  Change in total cholesterol, triglycerides, HDL, LDL and VLDL levels (mg/dl) will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Jehangir Hospital, Pune, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No